CLINICAL TRIAL: NCT03280862
Title: Does Targeted LV Lead Positioning Towards Latest Local Electric Activation at CRT Implantation Reduce Incidence of the Combined Endpoint "Death or Non-planned Hospitalisation for Heart Failure (HF)" in Patients With HF and Prolonged QRS
Brief Title: DANISH-CRT - Does Electric Targeted LV Lead Positioning Improve Outcome in Patients With Heart Failure and Prolonged QRS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Gentofte University Hospital (Unknown)
Responsible Party: Principal Investigator, Jens Cosedis Nielsen, Professor, DMSc, PhD, FESC, FEHRA, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-330-16
Record Dates: First submitted 2017-06-08; First posted 2017-09-13 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Branch Block, Bundle
Keywords: Heart Failure; Branch Block; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Intervention Model Description: Double-blind randomised controlled trial. Patients are included and randomised 1:1 into two groups for implantation of either
  1. a CRT-D/P device with the LV lead positioned according to the latest electrical activation in the CS (intervention group) or
  2. a CRT-D/P device with the LV lead positioned preferentially in a posterolateral, non-apical position (control group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients are unaware of treatment arm. All patients undergo the same pre-implant program and follow-up. Healthcare personel performing follow-up are blinded for treatment arm. Outcome events are evaluated by a committee blinded for treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Implantation of a Cardiac Resynchronisation Therapy (CRT) pacing device with or without Implanted Cardioverter Defibrillator with the LV lead positioned preferentially in a posterolateral, non-apical position
  Interventions: Device: Implantation of a Cardiac Resynchronisation Therapy (CRT) pacing device with or without Implanted Cardioverter Defibrillator
- Intervention (Experimental): Implantation of a Cardiac Resynchronisation Therapy (CRT) pacing device with or without Implanted Cardioverter Defibrillator with the LV lead positioned according to the latest electrical activation in the CS
  Interventions: Device: Implantation of a Cardiac Resynchronisation Therapy (CRT) pacing device with or without Implanted Cardioverter Defibrillator

INTERVENTIONS:
Device: Implantation of a Cardiac Resynchronisation Therapy (CRT) pacing device with or without Implanted Cardioverter Defibrillator — Implantation of CRT-P/-D device

SUMMARY:
Heart failure is a leading cause of morbidity and mortality. Cardiac resynchronization therapy (CRT) is a well-established treatment for patients with symptomatic heart failure in spite of optimised medical treatment (OMT), reduced left ventricular pump function with left ventricular ejection fraction (LVEF) ≤ 35% and prolonged activation of the ventricles (bundle branch block: BBB). CRT is established by implanting an advanced pacemaker system with three leads in the right atrium, right ventricle, and in the coronary sinus (CS) for pacing the left ventricle (LV), and often is combined with an implantable defibrillator (ICD) function. On average, CRT treatment improves longevity, quality of life and functional class, and reduces heart failure symptoms. Thus, at present, CRT is indicated for heart failure patients on OMT with BBB or chronic right ventricular (RV) pacing.

It is, however, a significant problem that 30-40% of CRT patients do not benefit measurably - showing symptomatic improvement or improved cardiac pump function - from this therapy (socalled non-responders). LV lead placement is one of the major determinants of beneficial effect from CRT.

Observational studies and three randomised trials with small sample sizes indicate that targeted placement of the LV lead towards a late activated segment of the LV may be associated with improved outcome. Based on this literature, some physicians already search for late activation when positioning the LV lead. However, such a strategy was never tested in a controlled trial with a sample size sufficient to investigate important clinical outcomes. Detailed mapping for a late activation may increase operating times and infection risk, result in use of more electrodes and wires, thereby increasing costs, and increase radiation exposure for patient and staff. Placement of the LV lead in late activated areas close to myocardial scar may even result in higher risk of arrhythmia and death.

At present, it is completely unsettled whether targeted positioning of the LV lead to the latest electrically activated area of LV is superior to contemporary standard CRT with regard to improving prognosis for patients with heart failure and BBB.

The present study aims to test whether targeting the placement of the LV lead towards the latest electrically activated segment in the coronary sinus branches improves outcome as compared with standard LV lead implant in a patient population with heart failure and CRT indication.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure, NYHA II, III, outpatient IV
* LVEF ≤35% measured by echocardiography
* Optimal medical treatment for heart failure
* Bundle Branch Block
* Indication for primary CRT-D or CRT-P implantation or upgrade from RV pacing (pacemaker or ICD) to CRT-D or CRT-P
* Ischemic heart disease (IHD) or non-IHD
* Sinus rhythm or atrial fibrillation
* Life expectancy >2 years
* Signed informed consent

Exclusion Criteria:

* NYHA class I
* Acute mycardial infarction (AMI) within the latest 3 months
* Coronary artery bypass graft (CABG) within the latest 3 months
* Life expectancy <2 years
* Participation in another clinical trial of experimental treatment
* Contraindication for establishing implantable device treatment
* Previously implanted CRT system
* Does not wish to participate

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Death or first non-planned hospitalisation for heart failure | All patients will be followed until the last included patient has been followed for two years
  Time to death or first non-planned hospitalisation for heart failure

SECONDARY OUTCOMES:
Death | All patients will be followed until the last included patient has been followed for two years
  Time to death
Non-planned hospitalisation for heart failure | All patients will be followed until the last included patient has been followed for two years
  Time to first non-planned hospitalisation for heart failure
Sudden death | All patients will be followed until the last included patient has been followed for two years
  Time to sudden death
Cardiac death | All patients will be followed until the last included patient has been followed for two years
  Time to cardiac death
Clinical response | Follow-up at 3, 6, 12, 24 and 48 months
  Increase in New York Heart Association (NYHA) class (≥1 class from baseline) or improved walking distance by six-minute walk test (6MWT) (≥10% from baseline)
Quality of Life (QoL) | Follow-up at 6, 12, 24 and 48 months
  Changes in score from baseline to follow-up
Patient Reported Outcomes (PROs) | Follow-up at 6, 12, 24 and 48 months
  Changes in score from baseline to follow-up
Echocardiographic measures of LV function | Follow-up at 6, 12, 24 and 48 months
  Changes from baseline to follow-up in left ventricular ejection fraction (%)
Time to first appropriate ICD Therapy | All patients will be followed until the last included patient has been followed for two years
  Time to first appropriate ICD therapy (antitachycardia pacing (ATP) or shock therapy)
Time to first inappropriate ICD Therapy | All patients will be followed until the last included patient has been followed for two years
  Time to first inappropriate ICD therapy (antitachycardia pacing (ATP) or shock therapy)
Numbers of appropriate ICD Therapies | All patients will be followed until the last included patient has been followed for two years
  Numbers of appropriate ICD therapies (antitachycardia pacing (ATP) or shock therapy)
Numbers of inappropriate ICD Therapies | All patients will be followed until the last included patient has been followed for two years
  Numbers of inappropriate ICD therapies (antitachycardia pacing (ATP) or shock therapy)
Ventricular tachycardia (VT)/ventricular fibrillation (VF) | All patients will be followed until the last included patient has been followed for two years
  Time to first episode of VT/VF
Persistent atrial fibrillation | All patients will be followed until the last included patient has been followed for two years
  Recorded by the implanted device
Any atrial fibrillation | All patients will be followed until the last included patient has been followed for two years
  >30 seconds recorded by the implanted device
Implantation time | 0-6 hours, assessed at completion of implantation procedure
  Procedure time at implantation
Fluoroscopy time | 0-120 minutes, assessed at completion of implantation procedure
  Fluoroscopy time at implantation in minutes
Fluoroscopy dose | Assessed <24 hours after implantation initiation
  Fluoroscopy dose at implantation in mGy
Equipment used at implantation | Assessed <24 hours after implantation initiation
  Number of LV leads (0-5) used at implantation
Device-related outcomes | All patients will be followed until the last included patient has been followed for two years
  Periprocedural: lead re-operation, pneumothorax, hemothorax, pericardial bleeding/tamponade and later (30 days post implantation): LV lead re-operation, device replacement due to battery depletion, and infection requiring extraction
Battery replacements | All patients will be followed until the last included patient has been followed for two years
  Number of device replacements during the study period due to battery depletion
Battery longevity estimate | All patients will be followed until the last included patient has been followed for two years
  Measured by actual device battery longevity + estimated remaining device battery longevity as reported by the device at last study follow-up
QRS complex width | All patients will be followed until the last included patient has been followed for two years
  Changes in the ECG parameter QRS complex width during follow-up
QRS complex morphology | All patients will be followed until the last included patient has been followed for two years
  Changes in the ECG parameter QRS complex morphology during follow-up
Predictive value of P-wave | All patients will be followed until the last included patient has been followed for two years
  Predictive value of the baseline ECG parameter P-wave on clinical outcome measures in the entire cohort and between the two treatment groups
Predictive value of QRS complex width | All patients will be followed until the last included patient has been followed for two years
  Predictive value of the baseline ECG parameter QRS complex width on clinical outcome measures in the entire cohort and between the two treatment groups
Predictive value of QRS complex morphology | All patients will be followed until the last included patient has been followed for two years
  Predictive value of the baseline ECG parameter QRS complex morphology on clinical outcome measures in the entire cohort and between the two treatment groups
Changes in cardiac chamber dimensions | All patients will be followed until the last included patient has been followed for two years
  Volumes of cardiac chambers (left ventricle, left atrium, right ventricle, right atrium) measured by echocardiography and cardiac CT during follow-up in the entire cohort and between the two treatment groups
Changes in left ventricular ejection fraction LVEF | All patients will be followed until the last included patient has been followed for two years
  Changes in cardiac chamber function measured by echocardiography and cardiac CT during follow-up in the entire cohort and between the two treatment groups
Changes in right ventricular ejection fraction RVEF | All patients will be followed until the last included patient has been followed for two years
  Changes in cardiac chamber function measured by echocardiography and cardiac CT during follow-up in the entire cohort and between the two treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Jens C Nielsen, Principal Investigator — Aarhus University Hospital
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Gentofte University Hospital, Gentofte Municipality
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kronborg MB, Frausing MHJP, Svendsen JH, Johansen JB, Riahi S, Haarbo J, Poulsen SH, Eiskjaer H, Kober L, Ovrehus K, Sommer AM, Schou M, Norgaard BL, Risum N, Poulsen MK, Sogaard P, Sandgaard N, Kofoed KF, Hansen TF, Graff C, Pedersen SS, Skals RG, Nielsen JC. Does targeted positioning of the left ventricular pacing lead towards the latest local electrical activation in cardiac resynchronization therapy reduce the incidence of death or hospitalization for heart failure? Am Heart J. 2023 Sep;263:112-122. doi: 10.1016/j.ahj.2023.05.011. Epub 2023 May 21. PMID 37220821